CLINICAL TRIAL: NCT05618275
Title: Role of Neutralizing Antibodies in the Prediction and Treatment of BK Virus Infection in Hematopoietic Stem Cell Allograft Patients at the Pediatric Oncology-hematology Department of the University Hospital of Strasbourg (HUS)
Brief Title: Role of Neutralizing Antibodies in the Prediction and Treatment of BK Virus Infection in Hematopoietic Stem Cell Allograft Patients at the Pediatric Oncology-hematology Department of the HUS
Acronym: BKV-Allograf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7635
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: BK Virus Infection
Keywords: BK virus infection; Neutralizing antibodies; Hematopoietic stem cell; Polyomaviridae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BK virus (BKV) belongs to the Polyomaviridae family. The primary infection, generally asymptomatic, occurs during childhood. The virus then persists in latent form in the body, mainly in the epithelial cells of the kidney and urinary tract. Cellular immunosuppression favors BKV replication. It is responsible for pathologies of the renal-urinary tract such as BKV-associated nephropathy (BKVAN) in kidney transplant recipients, hemorrhagic cystitis (HC) in hematopoietic stem cell (HSC) recipients or ureteral stenosis.

To date, there is no specific antiviral treatment against BKV. The management of patients is essentially symptomatic and requires a multidisciplinary approach. It is therefore necessary to identify early prognostic markers for the occurrence of CH and to develop new therapeutic strategies.

ELIGIBILITY:
Inclusion criteria:

* Adult patient aged 18 to 19 years
* Minor patient (from birth to 17 years old)
* HSC allograft patient managed by the pediatric oncology-hematology service of the HUS, between 01/01/2015 and 31/12/2019

Exclusion Criteria:

* Opposition of the patient (or parental authority holders) to participate in the study
* Biological resources from a patient who does not meet all inclusion criteria
* Patient deprived of liberty or under court protection
* Patient under guardianship or curatorship

Ages: 1 Year to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: HSC allograft patient managed by the pediatric oncology-hematology service of the HUS, between 01/01/2015 and 31/12/2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the role of anti-BKV neutralizing antibodies in HSCT patients in the pediatric oncology-hematology department of the HUS | Files analysed retrospectively from January 01, 2015 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service Laboratoire de Virologie - PTM - CHU de Strasbourg - France, Strasbourg, France